CLINICAL TRIAL: NCT03318744
Title: Antiplatelet Therapy in Secondary Prevention for Patient With Silent Brain Infarction
Brief Title: Antiplatelet Therapy for Silent Brain Infarction
Acronym: ANTISBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Shenyang (Other)
Responsible Party: Principal Investigator, Dr. Yi Sui, Director of Neurology, First People's Hospital of Shenyang
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FirstPHShenyang
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Brain Infarction
Keywords: Silent Brain Infarction; Antithrombotics; Antiplatelet; Aspirin; Asymptomatic
MeSH Terms: conditions — Brain Infarction | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin 100mg (Experimental): Participants will be given aspirin 100mg once per day.
  Interventions: Drug: Aspirin
- placebo (Placebo Comparator): Participants will be given placebo oral tablets once per day.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Aspirin — Aspirin is one of the most widely used antithrombotic agents to prevent recurrent ischemic stroke for patients with prior symptomatic ischemic stroke.
  Other Names: Bayaspirin
  Arms: aspirin 100mg
Drug: Placebo Oral Tablet — Placebo resembling aspirin tablet will be be given to participants in control arm.
  Arms: placebo

SUMMARY:
Silent brain infarction (SBI) or incidental infarct is common. Recent studies revealed individuals with SBI have an increased risk of future stroke. Even though the 2014 AHA/ASA recommendation for ischemic stroke and transient ischemic attack considered SBI as an entry point for secondary prevention, convincing evidence with regard to the preventive efficacy of antiplatelet therapy against incident stroke in SBI is scant. Investigators examine if antiplatelet therapy can effectively decrease the incidence of future stroke in SBI individuals.

DETAILED DESCRIPTION:
SBI is defined as a focal hyperintense lesion on T2-weighted images and/or fluid-attenuated inversion recovery with no corresponding symptoms in the clinical history of the patient that could be attributed to the lesion. SBI were distinguished from nonspecific subcortical and periventricular white matter lesions by the presence of a corresponding hypointense lesion on T1-weighted images.

The prevalence of SBI varies from 5% to 62% in healthy population. To date, few studies investigate the association between SBI and ethnicity. The effectiveness of antithrombotics including aspirin against future symptomatic stroke in SBI patients remains to be established. Due to the high prevalence of ICAS among Chinese, and its nature of artery-to-artery microembolisms, investigators hypothesize that the prevalence of SBI among Chinese might be significantly higher than other races such as Caucasians and African-Americans.

Recent study has revealed that SBI is associated with an 2-fold increase of future ischemic stroke. Yet, interventions such as antiplatelet therapies for reducing the stroke risk in SBI patients have not been investigated to our best knowledge. In this study, investigators examine whether regular oral aspirin can reduce the incidence of cerebrovascular events and mortality in SBI patients.

ELIGIBILITY:
Inclusion Criteria:

* cerebral infarction(s) identified by CT/MRI (≥ 3mm in diameter)
* absence of signs or symptoms of neurological dysfunction ascribed to the lesion(s)
* absence of PMH of neurological dysfunctions due to CNS lesion(s)

Exclusion Criteria:

* Age under 45 years or above 80 years
* PMH of ICH within 180 days
* PMH of lobar hemorrhage of anytime
* Neuroimaging evidence suggesting cerebral microbleeds
* High risk of bleeding (e.g. recurrent gastrointestinal or genitourinary bleeding, active peptic ulcer disease)
* Anticipated requirement for long-term use (more than 28 days) of anticoagulants (e.g. recurrent deep vein thrombosis)
* Prior long-term use of anticoagulants (more than 28 days) or antiplatelet agents (more than 28 days)
* Prior retinal stroke/TIA (diagnosed either clinically or by imaging)
* Intolerance or contraindications to aspirin (including thrombocytopenia, prolonged INR)
* Prior ipsilateral carotid endarterectomy/stent
* Stenosis of culprit artery ≥ 70% (detected by ultrasound, MRA, CTA or DSA)
* Atrial fibrillation, or acute myocardial infarction, or acute congestive heart failure
* Impaired renal function: glomerular filtration rate<60
* Mini Mental Status Examination score<24 (adjusted for age and education)
* Medical contraindication to MRI
* Pregnancy or women of child-bearing potential who are not following an effective method of contraception
* Unable or unwilling to provide informed consent
* Unlikely to be compliant with therapy/unwilling to return for frequent clinic visits
* Patients concurrently participating in another study with an investigational drug or device
* Independence ascribed to limb deformity or prior disability
* Acute myocardial infarction
* Acute congestive heart failure
* Other anticipated reasons for future application of antiplatelet agents other than aspirin (eg. recent stenting, interventional surgeries, Lower-Extremity Atherosclerotic Arterial Disease etc)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
composite outcome with any incident stroke, myocardial infarction and all-cause death | 24 months

SECONDARY OUTCOMES:
ischemic stroke, intracranial cerebral hemorrhage, any bleeding, independence (mRS≥2) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi Sui, MD PhD, Principal Investigator — First People's Hospital of Shenyang
Locations (1):
- Shenyang Brain Hsopital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Weber R, Weimar C, Wanke I, Moller-Hartmann C, Gizewski ER, Blatchford J, Hermansson K, Demchuk AM, Forsting M, Sacco RL, Saver JL, Warach S, Diener HC, Diehl A; PRoFESS Imaging Substudy Group. Risk of recurrent stroke in patients with silent brain infarction in the Prevention Regimen for Effectively Avoiding Second Strokes (PRoFESS) imaging substudy. Stroke. 2012 Feb;43(2):350-5. doi: 10.1161/STROKEAHA.111.631739. Epub 2012 Jan 19. PMID 22267825
- [Background] Chou CC, Lien LM, Chen WH, Wu MS, Lin SM, Chiu HC, Chiou HY, Bai CH. Adults with late stage 3 chronic kidney disease are at high risk for prevalent silent brain infarction: a population-based study. Stroke. 2011 Aug;42(8):2120-5. doi: 10.1161/STROKEAHA.110.597930. Epub 2011 Jun 23. PMID 21700935
- [Background] Nakagawa T, Sekizawa K, Nakajoh K, Tanji H, Arai H, Sasaki H. Silent cerebral infarction: a potential risk for pneumonia in the elderly. J Intern Med. 2000 Feb;247(2):255-9. doi: 10.1046/j.1365-2796.2000.00599.x. PMID 10692089
- [Background] Wang Y, Zhao X, Liu L, Soo YO, Pu Y, Pan Y, Wang Y, Zou X, Leung TW, Cai Y, Bai Q, Wu Y, Wang C, Pan X, Luo B, Wong KS; CICAS Study Group. Prevalence and outcomes of symptomatic intracranial large artery stenoses and occlusions in China: the Chinese Intracranial Atherosclerosis (CICAS) Study. Stroke. 2014 Mar;45(3):663-9. doi: 10.1161/STROKEAHA.113.003508. Epub 2014 Jan 30. PMID 24481975
- [Background] Caplan LR, Hennerici M. Impaired clearance of emboli (washout) is an important link between hypoperfusion, embolism, and ischemic stroke. Arch Neurol. 1998 Nov;55(11):1475-82. doi: 10.1001/archneur.55.11.1475. PMID 9823834
- [Background] Gupta A, Giambrone AE, Gialdini G, Finn C, Delgado D, Gutierrez J, Wright C, Beiser AS, Seshadri S, Pandya A, Kamel H. Silent Brain Infarction and Risk of Future Stroke: A Systematic Review and Meta-Analysis. Stroke. 2016 Mar;47(3):719-25. doi: 10.1161/STROKEAHA.115.011889. PMID 26888534
- [Background] Smith EE, Saposnik G, Biessels GJ, Doubal FN, Fornage M, Gorelick PB, Greenberg SM, Higashida RT, Kasner SE, Seshadri S; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Functional Genomics and Translational Biology; and Council on Hypertension. Prevention of Stroke in Patients With Silent Cerebrovascular Disease: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Feb;48(2):e44-e71. doi: 10.1161/STR.0000000000000116. Epub 2016 Dec 15. PMID 27980126